CLINICAL TRIAL: NCT06590649
Title: PILI 'Āina 2 Household Participants
Brief Title: Household Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PILI 'Āina 2 Household Members; R01HL168858 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes; Hypertension; Dyslipidemias; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Household Participants (Experimental): The household participants will be analyzed alongside the index participants to determine household-level effects from the intervention. Household participants must live in an index participant's household. Index participants are allowed to have up to 3 household participants.
  Interventions: Behavioral: Household-level effects

INTERVENTIONS:
Behavioral: Household-level effects — At 3 months, participants randomized to the PILI 'Āina intervention will receive a 6-month intervention centered around the use of a raised-bed home garden as the means of engaging household members to 1) increase their access to and intake of vegetables, 2) learn culturally relevant ways of preparing/cooking fresh vegetables through hands-on cooking lessons with local experts, and 3) build family cohesion through family bonding activities. Participants will be given all the equipment and materials (e.g., soil, seeds, instructions, setup of equipment) needed to grow their vegetables using their raised-bed home garden box throughout the entire study. They will receive seeds for the vegetables that can grow in a relatively short period (i.e., within 6 weeks). The household participants will be analyzed side by side with the index participants.
  Other Names: PILI 'Aina 2

SUMMARY:
Native Hawaiians' traditional lifestyles and diets ensured the mutual health and well-being of the land and its inhabitants, which stand in stark contrast to the disproportionately high prevalence of diet-related, cardiometabolic diseases they experience today. In this project, the investigators will adapt and test an evidence-based multilevel intervention entitled PILI 'Āina to improve the self-management of prevalent cardiometabolic diseases and reduce risk factors for developing new diet-related illnesses and implement and evaluate the impact and sustainability of community-wide cooking demonstrations. The objectives of this project are to optimize the effectiveness and sustainability of PILI 'Āina, improve diet quality, cardiometabolic markers, promote traditional Native Hawaiian diets, and improve social cohesion.

DETAILED DESCRIPTION:
The investigators will conduct a group-randomized controlled trial to test the effectiveness of PILI Aina for improving diet and health at the individual and household levels compared to a Diabetes Prevention Program Lifestyle Intervention only group. The investigators will enroll 180 Native Hawaiian adults with overweight or obesity and at least 1 other diet-related cardiometabolic condition (Type 2 diabetes, pre-diabetes, hypertension, pre-hypertension, dyslipidemia). These index participants will receive the 3-month educational program and then be randomized at the household level to the 6-month PILI Aina intervention or to a control group. Data collection will occur at baseline and 3, 9, and 12 months. Other adult household members will be invited to participate in data collection at the same time to evaluate household-level effects.

ELIGIBILITY:
Inclusion Criteria:

* Current resident of the household in which an index participant lives
* Willing to complete data collection protocols
* Fluent in written and spoken English

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Household Food Patterns | Month 3, Month 9, Month 12
  Household food patterns will be measured by 4 questions that assess the frequency of meal planning, eating meals with household members, bringing prepared restaurant foods home, and preparing meals with household members. The responses and scores range from 1- 1 day, 2- 2-3 days, 3- 4-5 days, 4- 6 days, 5- 7 days. Higher scores indicate greater household food patterns.
Food insecurity | Month 3, Month 9, Month 12
  Food insecurity will be measured by the 10-item Household Food Security Survey Module, which captures the qualitative and quantitative dimensions of household food supply, including psychological and behavioral responses of household members, and generates a binary indicator of food insecurity at the household level. The responses and scores range from 1-often true, 2-sometimes true, 3-never true. Higher scores indicate low food insecurity.
Nutrition Environment | Month 3, Month 9, Month 12
  The perceived 9-item nutrition environment will be measured by the Gustafson Perceived Nutrition Environment Measures questionnaire, which examines perceived access and availability of healthy foods within ~1 mile of the participant's home, and the availability and affordability of produce in the participant's primary food store. The responses and scores vary depending on the question including 0- disagree, 1-agree, and 0-not important, 1-slightly important, 2-moderately important, 3- important, 4-very important. Higher scores indicate higher perceived access and availability of food.
Physical Activity | Month 3, Month 9, Month 12
  The 3-item Physical Activity Questionnaire, which has been used with Native Hawaiians, will assess exercise frequency during the past month. It contains 3 items that assess moderate and vigorous exercise and changes in activity levels. The responses and scores vary depending on the question, including 0- rarely or never, 1- 2-3 times over the month, 2- about once a week, 3- 2-4 times a week, 4- more than 4 times a week. Higher scores indicate greater physical activity.

SECONDARY OUTCOMES:
Demographic Data- Date of Birth | Baseline
  Date of birth:
  * Month
  * Day
  * Year
Demographic Data- Biological Sex | Baseline
  Biological Sex:
  * Female
  * Male
Demographic Data- Marital status | Baseline
  Marital Status:
  * Never married
  * Currently married
  * Divorced or separated
  * Widow/widower
  * Domestic partnership/other
Demographic Data- Employment | Baseline
  Employment:
  * Full time
  * Part-time
  * Unemployed
  * Self-employed
  * Retired
  * Unable to work/other
  * Household caretaker
Demographic Data- Education | Baseline
  Education:
  * Less than high school
  * High school diploma/General Education Diploma (GED)
  * Some college/technical training
  * College degree
  * Graduate/professional degree
Demographic Data- Ethic Ancestry | Baseline
  Ethnic Ancestry:
  * Caucasian
  * Chinese
  * Filipino
  * Hawaiian
  * Latino
  * Japanese
  * Korean
  * Marshallese
  * Micronesian (specify)
  * Native American
  * Portuguese
  * Samoan
  * Other (specify)
Demographic Data- Household income | Baseline
  Household Income:
  * Under $49,999
  * $50,000-$74,999
  * $75,000-$99,999
  * $100,000-$124,999
  * Over $125,000
  Household income will be classified according to the US Census Bureau's poverty threshold by using a dichotomous variable. Participation in public assistance programs (e.g., Temporary Assistance for Needy Families, Supplemental Nutrition Assistance Program) will also be recorded.
Demographic Data- Household Composition | Baseline
  Household Composition:
  1. Who lives in your house full-time? (50% or more time spent in-house)
  * Parents
  * Children
  * Grandparents/great-grandparents
  * Other family members
    a. Of those people, what are their ages and genders?
  * Male: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Female: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
  * Number of other/non-binary: 17 years and under, 18-29 yrs, 30-39 yrs, 40-39 yrs, 50-59 yrs, 60+ yrs
Smoking/alcohol | Month 3, Month 9, Month 12
  Tobacco and alcohol use will be measured by using a measure developed by Dr. Kaholokula for PILI 'Ohana.
Neighborhood environment | Month 3, Month 9, Month 12
  Neighborhood environment will be measured by the 17-item modified Neighborhood Level Stressors Scale, which assesses participants' perceptions of 4 neighborhood dimensions (i.e., walkability, availability of healthy food, safety, and social cohesion). The responses and scores range from 1-strongly disagree, 2-somewhat disagree, 3- neutral, 4-somewhat agree, 5-strongly agree. Higher scores indicate low neighborhood level stressors.
Comorbidities | Month 3, Month 9, Month 12
  Existing comorbidities will be measured as whether the participant has ever been told by a healthcare professional that they have had a heart attack, heart failure, stroke, or chronic kidney disease.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kula no nā Po'e Hawai'i, Honolulu, Hawaii
  - Kapolei Community Development Corporation, Kapolei, Hawaii

IPD SHARING:
Plan to Share IPD: No